CLINICAL TRIAL: NCT00005334
Title: Effects of Personality and Context on Recovery From Coronary Artery Bypass
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4189; R01HL044436 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression

SUMMARY:
To study the personality and environmental factors that may determine the short-term and long-term sequelae of coronary artery bypass surgery (CABS).

DETAILED DESCRIPTION:
BACKGROUND:

Coronary artery bypass surgery, or CABS, is one of the most common surgical procedures for treating patients with coronary artery disease (CAD). A significant number of patients have accelerated atherosclerosis in the postsurgical period and require second and third operations. Moreover, relative to standard medical care, CABS does little to prolong life. The major benefit of the procedure is improving life quality. Thus, to enhance this major benefit of CABS, it is important to understand the factors, psychosocial as well as biological, that might enhance quality of life after CABS. The few available studies on the psychosocial aspects of recovery from CABS suggest that person variables evident prior to surgery are related to postsurgery quality of life. Of special interest here are gender, optimism, Type A, with its component behavior of hostility, and repressive style. The significance of these attributes derives from their theoretical and empirical relationships to the patient's illness representations and correspondent coping responses, and/or their relationship to risk for coronary heart disease (CHD). In addition to person variables, a number of environmental variables might also be expected to play a role in recovery. Variables such as socioeconomic status (SES), major life events, and quantity and quality of social support systems have all been shown to impact on health and illness. Moreover, from a slightly different perspective, the patient's illness itself can serve as an environmental variable impinging on the life of the person providing the primary support. Thus, it is also important to understand how the patient's illness impacts on the provider of the primary support.

DESIGN NARRATIVE:

A total of 305 patients between the ages of 25 and 70 scheduled for elective surgery at a major local hospital were evaluated two weeks prior to surgery on the day prior to surgery, and one week, six months, and two and a half years postsurgery. Primary support persons were evaluated three times--at intake, six months postsurgery, and two and a half years postsurgery. Medical information was obtained that permitted examination of the influences of psychosocial variables on recovery. Major personality variables under investigation were optimism, Type A, hostility, gender, repressive style, and to a lesser extent, anxiety, and neuroticism. Major environmental variables included quality and quantity of social support and availability of a primary support person. Main outcome variables for patients included satisfaction with different life domains, depression, return to work, normalization of life style, and new and recurrent morbidity. Main outcome variables for the support person included perceptions of burden, depression, and life satisfaction.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-07; Study Completion 1995-06 (Actual)

REFERENCES:
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Carver CS, Scheier MF. Situational coping and coping dispositions in a stressful transaction. J Pers Soc Psychol. 1994 Jan;66(1):184-95. doi: 10.1037//0022-3514.66.1.184. PMID 8126648
- [Background] Carver CS, Pozo C, Harris SD, Noriega V, Scheier MF, Robinson DS, Ketcham AS, Moffat FL Jr, Clark KC. How coping mediates the effect of optimism on distress: a study of women with early stage breast cancer. J Pers Soc Psychol. 1993 Aug;65(2):375-90. doi: 10.1037//0022-3514.65.2.375. PMID 8366426
- [Background] Newsom JT, Schulz R. Social support as a mediator in the relation between functional status and quality of life in older adults. Psychol Aging. 1996 Mar;11(1):34-44. doi: 10.1037/0882-7974.11.1.34. PMID 8726368
- [Background] Scheier MF, Bridges MW. Person variables and health: personality predispositions and acute psychological states as shared determinants for disease. Psychosom Med. 1995 May-Jun;57(3):255-68. doi: 10.1097/00006842-199505000-00007. PMID 7652126
- [Background] Scheier MF, Matthews KA, Owens JF, Schulz R, Bridges MW, Magovern GJ, Carver CS. Optimism and rehospitalization after coronary artery bypass graft surgery. Arch Intern Med. 1999 Apr 26;159(8):829-35. doi: 10.1001/archinte.159.8.829. PMID 10219928
- [Background] Nieboer AP, Schulz R, Matthews KA, Scheier MF, Ormel J, Lindenberg SM. Spousal caregivers' activity restriction and depression: a model for changes over time. Soc Sci Med. 1998 Nov;47(9):1361-71. doi: 10.1016/s0277-9536(98)00214-7. PMID 9783879